CLINICAL TRIAL: NCT03666416
Title: Acute Effects of Exercise in College Students With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Cynthia M Hartung, PhD, Associate Professor, University of Wyoming
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170220PL01463
Record Dates: First submitted 2018-08-31; First posted 2018-09-11 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Effects of; Exertion; Working Memory; Change in Sustained Attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a within-subjects design where participants complete outcome measures with and without exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sprint Interval Training (Experimental): Participants will be scheduled for two in-lab experimental appointments: sprint interval training (SIT) and Non-SIT. During the SIT appointment, the researcher will lead the participant through a set of stretches and three minutes of low-intensity cycling on a Schwinn AD2 Airdyne leg-cycling and arm-cranking ergometer to warm up and increase blood flow to active muscles. Participants will then complete 16 minutes of SIT, consisting of eight bouts of 20 seconds of cycling followed by 100 seconds of rest. Participants will complete computer-based tests of sustained attention and working memory during both the SIT (15 minutes following the exercise) and Non-SIT appointments.
  Interventions: Behavioral: Sprint Interval Training

INTERVENTIONS:
Behavioral: Sprint Interval Training — Participants will attend two experimental appointments, during which they will complete two identical executive functioning tasks (i.e., sustained attention, working memory). During one appointment, participants will receive the sprint interval training manipulation prior to completing the tasks.

SUMMARY:
The overall objective of this study is to examine physical exercise as an intervention for ADHD. The rationale for the proposed study is that physical exercise could serve as an effective treatment for college students with ADHD that has low costs, low risks, and ancillary health benefits and may address the limitations of existing treatments. The central hypothesis is that college students with ADHD will exhibit greater degrees of improvement in executive functioning (i.e., sustained attention, working memory) immediately following sprint interval training (SIT), relative to non-ADHD peers. This hypothesis was formulated based on preliminary studies demonstrating reduced ADHD symptoms and improved executive functioning following physical exercise. Multiple 2 (ADHD vs. control) x 2 (male vs. female) x 2 (exercise vs. none) repeated measures ANOVAs will be conducted to compare students with ADHD (n = 24) to controls (n = 24).

The expected outcomes are to confirm this hypothesis and demonstrate the need for further study of physical exercise. If confirmed, the results will provide pilot data for a larger NIH grant proposal aimed at further examining the acute effects of physical exercise (i.e., improved cognitive functioning immediately following exercise) and also the chronic effects of physical exercise (i.e., improved functioning after engaging in regular exercise for an extended period). This outcome is expected to have an important positive impact because physical exercise may serve as an effective treatment for college students with ADHD that is less risky than stimulants, less time-consuming than therapy, and provides ancillary health benefits (i.e., increasing physical fitness, decreasing obesity).

DETAILED DESCRIPTION:
Participant enrollment will consist of forty-eight University of Wyoming (UW) and Laramie County Community College (LCCC) students (24 ADHD group, 24 comparison group) with an even distribution of men and women in each group. Power analyses (G*Power 3.1) indicated a sample of at least this size is needed to provide 80% power to detect medium effects which have been observed in samples of children with ADHD. Students taking medications that may confound cognitive performance (e.g., antipsychotics, sedatives), are outside the age range (18-25 years), or are at an elevated risk for physical exercise contraindications will be excluded. Prospective ADHD group participants will be recruited through four means. First, students who complete a separate study and endorse five or more inattention (IA) symptoms or report being previously diagnosed with ADHD will be invited for an eligibility assessment. Second, recruitment flyers will be posted on campus. Third, participants will be contacted from previous studies who were diagnosed with ADHD and consented to contact for future research. Fourth, university medical and mental health staff will advertise the study to student clients who have ADHD. Comparison group subjects will be composed of students who complete a separate study, who disavow being diagnosed with ADHD, and endorse three or fewer IA symptoms. As students enroll in the ADHD group, age- and sex-matched comparison subjects will be enrolled. Prior to study enrollment, prospective participants must stratify as being at low risk for physical exercise contraindications using a health history screening questionnaire. Prospective ADHD participants must also meet diagnostic criteria for ADHD on a structured clinical interview.

All prospective participants will attend an in-lab appointment to confirm their eligibility, including (a) stratifying as being at low risk for physical exercise contraindications and (b) ADHD prospects meeting diagnostic threshold. After enrolling in the study, participants will be scheduled for two in-lab experimental appointments: sprint interval training (SIT) and Non-SIT. The ordering of experimental appointments will be counterbalanced. This will be done to evaluate possible appointment ordering effects and minimize confounding effects. Both appointments will be scheduled in the mornings, on the same day of the week and at the same time of day. Participants will be asked to wear athletic clothing, as well as abstain from exercise, alcohol, caffeine, and stimulant medication for 12 hours prior to their experimental appointments to minimize the influence they may have on our independent (exercise) and dependent variables (executive functioning). Participants will complete the execute functioning tasks (i.e., Continuous Performance Task or CPT, Digit Span, Letter-Number Sequencing, and Spatial Span or SS) during both the Non-SIT and SIT appointments. They will also be sent a modified mood (i.e., Depression, Anxiety, and Stress Scale or DASS) and ADHD symptoms (Barkley Adult ADHD Rating Scale or BAARS) questionnaire the morning following all experimental appointments. High-intensity SIT was chosen for the proposed study because moderate- to high-intensity aerobic exercises appears to lead to the greatest improvements in cognitive performance among youth with ADHD. The researcher will lead the participant through a set of stretches and 3 minutes of low-intensity cycling on a Schwinn AD2 Airdyne leg-cycling and arm-cranking ergometer to warm up and increase blood flow to active muscles. Participants will then complete 16 minutes of SIT, consisting of eight bouts of 20 seconds of cycling followed by 100 seconds of rest. After each interval, participants will be asked to provide their perceived exertion during the interval, and the researcher will record participant's peak interval heart rate (HR). These measurements are taken to validate that participants exercised at a high intensity. The experimenter will provide encouragement to the participant to work towards ≥85% of their maximum HR. After the eighth and last interval, the participant will rest for 15 minutes before completing the cognitive tasks (i.e., CPT, Digit Span, Letter-Number Sequencing, and SS).

Prior to analyses, all variables will be screened. Violations of statistical assumptions will be addressed through data transformations or nonparametric statistics. Relative improvements on objective measurements of EF (i.e., CPT, Digit Span, Letter-Number Sequencing, and SS performance indices) will be examined through 2 (ADHD vs. comparison) x 2 (men vs. women) x 2 (Non-SIT vs. SIT) repeated measures ANOVAs. When interaction effects are significant, paired samples t-tests will be used to evaluate group differences. When interaction effects fail to reach statistical significance, independent samples t-tests will be used to evaluate group differences. The magnitude of omnibus effects for repeated measures ANOVAs will be calculated using partial eta-squared (ηp2). Within-group effects (Cohen's d) and corresponding confidence intervals for within-group effect sizes will be standardized using the variability of non-SIT scores. Between-group effects will be calculated using Hedges g. Values for ηp2 of .01, .06, and .14 will be considered small, medium, and large effects, respectively; corresponding values for d and g are .20, .50, and .80.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 29 years.
* University of Wyoming (UW) or Laramie County Community College (LCCC) student.

Exclusion Criteria:

* Predominantly hyperactive/impulsive presentations of ADHD (ADHD-HI), as this presentation is unusual in adulthood.
* Use of medications that negatively affect cognitive performance (e.g., sedatives, antipsychotics).
* Pregnancy or trying to become pregnant.
* Non-ambulatory or relying on walking aids for ambulation.
* History of a stroke or an aneurysm.
* High risk for physical exercise contraindications due to genetic/medical conditions (e.g., cardiovascular or pulmonary disease).
* Exercise or physical activity restrictions imposed by a health provider.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Continuous Performance Test (CPT) from appointment 1 to 2 | Completed at each experimental appointment over a period of two weeks
  The CPT is a standardized computer-administered test consisting of four-digit numbers that are presented for 200ms on a white screen with 1500ms between the presentation of each number. Participants must press the spacebar as quickly as possible when the preceding four-digit number matches the current four-digit number Participants will complete the CPT as a measure of sustained attention at each experimental appointment. For the SIT appointment, participants will complete the CPT 15 minutes after exercise termination.
Change in Digit Span from appointment 1 to 2 | Completed at each experimental appointment over a period of two weeks
  The Digit Span (Wechsler, 2008) subtest of the Wechsler Adult Intelligence Scale (WAIS-IV) is an auditory working memory task. The researcher will say numbers aloud at a rate of one number per second. The participant will be tasked with remembering and repeating the numbers in a prescribed (forward, backward, sequencing) order. Participants will complete the Digit Span (forward, backward and sequencing) auditory working memory task at each experimental appointment. For the SIT appointment, participants will complete the Digit Span (forward, backward and sequencing) tasks approximately 15 minutes after exercise termination.
Change in Letter-Number Sequencing from appointment 1 to 2 | Completed at each experimental appointment over a period of two weeks
  The Letter-Number Sequencing (Wechsler, 2008) task is a supplemental subtest of the Wechsler Adult Intelligence Scale (WAIS-IV) that measures auditory working memory. Researchers will read a sequence of letters and numbers, and the participant will attempt to recall the numbers in ascending order and the letters in alphabetical order. Participants will complete the Letter-Number Sequencing auditory working memory task at each experimental appointment. For the SIT appointment, participants will complete the Letter-Number Sequencing task approximately 15 minutes after exercise termination.
Change in Spatial Span (SS) from appointment 1 to 2 | Completed at each experimental appointment over a period of two weeks
  The Spatial Span (SS) is a computer-administered task assessing visuospatial working memory. Participants will be tasked with remembering the order of stimuli that are presented in forward and backward sequences. Participants will complete the SS visuospatial working memory task at each experimental appointment. For the SIT appointment, participants will complete the SS task approximately 15 minutes after exercise termination.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale-Modified (DASS-M) | Completed the day after each experimental appointment over a period of two weeks
  This scale includes 21 questions to measure current mood and stress levels. Items include a choice of four responses from "Did not apply to me at all," to "Applied to me very much." Participants will receive the survey via text and email the morning after their experimental appointment. They will be instructed to complete the DASS-M regarding their emotional experiences of depression, anxiety, and stress from "yesterday (from the time after your lab appointment until you went to bed)."
Barkley Adult ADHD Rating Scale-Modified (BAARS-M) | Completed the day after each experimental appointment over a period of two weeks
  The BAARS includes 18 items that closely follow the Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-5; APA, 2013) criteria for ADHD. Participants will be asked to rate their current behavior over the past 6 months from 0 (Never/Rarely) to 3 (Very Often).Participants will receive the survey via text and email the morning after their experimental appointment. They will be instructed to complete the BAARS-M regarding their ADHD-related behavior from "the previous day."

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Hartung, Ph.D., Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoza B, Smith AL, Shoulberg EK, Linnea KS, Dorsch TE, Blazo JA, Alerding CM, McCabe GP. A randomized trial examining the effects of aerobic physical activity on attention-deficit/hyperactivity disorder symptoms in young children. J Abnorm Child Psychol. 2015 May;43(4):655-67. doi: 10.1007/s10802-014-9929-y. PMID 25201345
- [Background] Chang YK, Liu S, Yu HH, Lee YH. Effect of acute exercise on executive function in children with attention deficit hyperactivity disorder. Arch Clin Neuropsychol. 2012 Mar;27(2):225-37. doi: 10.1093/arclin/acr094. Epub 2012 Feb 3. PMID 22306962
- [Background] Choi JW, Han DH, Kang KD, Jung HY, Renshaw PF. Aerobic exercise and attention deficit hyperactivity disorder: brain research. Med Sci Sports Exerc. 2015 Jan;47(1):33-9. doi: 10.1249/MSS.0000000000000373. PMID 24824770
- [Background] Neudecker C, Mewes N, Reimers AK, Woll A. Exercise Interventions in Children and Adolescents With ADHD: A Systematic Review. J Atten Disord. 2019 Feb;23(4):307-324. doi: 10.1177/1087054715584053. Epub 2015 May 11. PMID 25964449
- [Background] Gapin, J. I., Labban, J. D., Bohall, S. C., Wooten, J. S., & Chang, Y. (2015). Acute exercise is associated with specific executive functions in college students with ADHD: A preliminary study. Journal of Sport and Health Science, 4, 89-96. doi:10.1016/j.jshs.2014.11.003
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Borg, G. A. (1998). Borg's perceived exertion and pain scales. Champaign, IL: Human Kinetics.
- [Background] Howell, D. C. (2011). Confidence intervals on effect size. http://www.uvm.edu/~dhowell/methods8/Supplements/Confidence%20Intervals%20on%20Effect%20Size.pdf. Accessed August 23, 2013.
- [Background] Hedges, L. V. (1982). Fitting categorical models to effect sizes from a series of experiments. Journal of Educational Statistics, 7, 119-37. doi: 10.2307/1164961
- [Background] Cohen, J. (1988). Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ: Lawrence Erlbaum.